CLINICAL TRIAL: NCT05693142
Title: A Phase 1/2/3 Open-label Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacodynamics, and Pharmacokinetics of Intravenous RGX-202 Gene Therapy in Males With Duchenne Muscular Dystrophy (DMD)
Brief Title: AFFINITY DUCHENNE: RGX-202 Gene Therapy in Participants With Duchenne Muscular Dystrophy (DMD)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGX-202-1101
Record Dates: First submitted 2023-01-04; First posted 2023-01-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Gene therapy; DMD; Duchenne Muscular Dystrophy; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Dose Evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Cohort 1 and 1b: RGX-202 Dose 1 (Experimental): A single IV infusion of RGX-202 at a dose of 1×10^14 GC/kg body weight
  Interventions: Genetic: RGX-202
- Part 1: Cohort 2, 2c;, and Part 2; and Part 3: RGX-202 Dose 2 (Experimental): A single IV infusion of RGX-202 at a dose of 2x10^14 GC/kg body weight
  Interventions: Genetic: RGX-202

INTERVENTIONS:
Genetic: RGX-202 — RGX-202 is a recombinant AAV8 containing a transgene encoding a novel microdystrophin

SUMMARY:
RGX-202 is a gene therapy designed to deliver a transgene for a novel microdystrophin that includes functional elements of naturally-occurring dystrophin including the C-Terminal (CT) domain.

This is a multicenter, open-label dose evaluation clinical study to assess the safety, tolerability, and clinical efficacy of a one-time intravenous (IV) dose of RGX-202 in participants with Duchenne.

For additional information on how to participate (or be considered for the study), please follow this link: https://mytomorro.ws/affinity-ct-gov

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (Duchenne) is a rare genetic disorder, caused by mutations in the gene responsible for making dystrophin, a protein of central importance for muscle cell structure and function. The absence of functional dystrophin protein in individuals with Duchenne results in cell damage during muscle contraction leading to cell death, inflammation, and fibrosis in muscle tissues, and ultimately progressive muscle weakness. RGX-202 is designed to use the AAV8 vector to deliver a transgene to muscle cells that encodes a novel microdystrophin that includes the functional elements of naturally occurring dystrophin including the C-Terminal (CT) domain.

This is a multicenter, phase I/II/III, open-label study to evaluate the safety, tolerability, pharmacodynamics (microdystrophin protein levels), pharmacokinetic, and clinical efficacy of RGX-202 when administered IV as one-time dose to ambulant male participants with Duchenne. A comprehensive, short-term, prophylactic immunosuppression regimen will be administered during treatment to mitigate a potential immune response. This study is being conducted in three sequential parts: a phase I/II study (Part 1), a phase 3 pivotal study (Part 2) and a confirmatory study (Part 3). Part 1 will study a one-time dose of RGX-202 (1x10^14 or 2x10^14 GC/kg) in up to 15 participants with Duchenne. In part 1, the primary objective is to evaluate the safety and tolerability of RGX-202 through 52 weeks. Part 2 (Pivotal Expansion) will study a single dose of RGX-202 (2x10^14 GC/kg) in approximately 30 participants. After the last Part 2 participant is dosed, enrollment into the confirmatory study (Part 3) will be initiated. The target enrollment for the confirmatory study (Part 3) is approximately 30 participants. Participants will be assessed at various time points for 104 weeks after receiving RGX-202. All participants will be given the opportunity to enroll in a separate long-term follow-study in accordance with the US federal government guidelines for the safety follow-up of patients receiving gene therapy.

ELIGIBILITY:
Part 1 - Key Inclusion Criteria:

* The participant's legal guardian(s) is (are) willing and able to provide written, signed informed consent prior to any study-related procedures; and, where applicable, the minor participant has provided written or verbal assent according to local requirements.
* Is a male at least 4 years of age and less than 12 years of age at consent or 1 to <4 years of age at the time of dosing and ≥ 10 kg at the time of screening.
* Must meet any of the following criteria:

  * DMD gene mutation in exons 18 and above, and a clinical picture consistent with typical DMD with the exception of a participant (Cohort 1b) with DMD gene mutation in exons 12-17.
  * Participant is able to walk 100 meters independently without assistive devices. Cohort 2c participant must be able to walk 10 meters independently without assistive devices. Cohort 1b participant must be able to walk with or without assistive devices.
  * Participant is able to complete the TTSTAND per protocol-specific criteria.
  * Participant has been on a stable dose of systemic glucocorticoids according to the standard of care for at least 12 weeks. Cohort 2c participants must be consistently on or off a stable dose of systemic glucocorticoids according to the standard of care for at least 12 weeks.
  * Clinical laboratory test results, including hepatic and renal function, are within the normal range during screening, or if abnormal, are not clinically significant, in the opinion of the investigator.
  * Documentation is provided at screening visit for participant's adherence to the local country's vaccination schedule. The parent(s) or legal guardian(s) must be willing to have their child receive a meningococcal vaccine, if not already vaccinated.
  * Participant and parent(s)/legal guardian(s) are willing and able to comply with scheduled visits, study intervention administration plan, and study procedures.

Part 2 and 3 Inclusion Criteria:

* The participant's legal guardian(s) is (are) willing and able to provide written, signed informed consent prior to any study-related procedures; and, where applicable, the minor participant has provided written or verbal assent according to local requirements.
* DMD gene mutation with any mutation except for those with deletions or point mutations in exons 8, 9 and/or 10.
* Participant is able to complete the TTSTAND per protocol-specific criteria.
* Clinical laboratory test results, including hepatic and renal function, are within the normal range during screening, or if abnormal, are not clinically significant, in the opinion of the investigator.
* Documentation is provided at screening visit for participant's adherence to the local country's vaccination schedule. The parent(s) or legal guardian(s) must be willing to have their child receive a meningococcal vaccine, if not already vaccinated.
* Participant and parent(s)/legal guardian(s) are willing and able to comply with scheduled visits, study intervention administration plan, and study procedures.
* Is a male at least 1 year of age and ≥ 10 kg at the time of screening.
* Participants 1 to <4 years of age must meet the following criteria:

  * is able to walk 10 meters independently without assistive devices.
  * must be consistently on or off a stable dose of systemic glucocorticoids according to the standard of care for at least 12 weeks.
* Participants 4 years and older must meet the following criteria:

  * are able to walk 100 meters independently without assistive devices.
  * have been on a stable dose of systemic glucocorticoids according to the standard of care for at least 12 weeks.
  * have a NSAA total score ≥16.

Part 1 Exclusion Criteria:

* Participant has any condition that would contraindicate treatment with immunosuppression.
* Participant has received ataluren (a protein restoration therapy) or an exon-skipping therapy for the treatment of DMD within 6 months of study entry or is unable to refrain from taking ataluren or exon-skipping therapy for a duration of 5 years from the time of RGX-202 administration.
* Participant has received any investigational or commercial gene therapy product over his lifetime.
* Participant is currently taking any other investigational intervention (other than corticosteroids) or has taken any other investigational intervention (other than corticosteroids) within 3 months prior to the scheduled Day 1 intervention. If your corticosteroid is vamorolone, the participant will be asked to temporarily convert his daily dosing to prednisolone/prednisone during a short period of time around RGX-202 administration. He will be allowed to revert back to his baseline vamorolone regimen at the original per kilogram dose at which he entered the study and should remain on this for 24 months unless the investigator determines that this is not clinically indicated or possible.
* Participant has impaired cardiac function defined as a left ventricular ejection fraction of < 55% on screening cardiac assessments (echocardiogram or MRI).
* Participant is not a good candidate for the study, in the opinion of the investigator.

Part 2 and 3 Exclusion Criteria:

* Participant has any condition that would contraindicate treatment with immunosuppression.
* Participant has received givinostat within 3 months of study entry or has received ataluren (a protein restoration therapy) or an exon-skipping therapy for the treatment of DMD within 6 months of study entry or is unable to refrain from taking ataluren or exon-skipping therapy for a duration of 5 years from the time of RGX-202 administration.
* Participant has received any investigational or commercial gene therapy product over his lifetime.
* Participant is currently taking any other investigational intervention (other than corticosteroids) or has taken any other investigational intervention (other than corticosteroids) within 3 months prior to the scheduled Day 1 intervention. If your corticosteroid is vamorolone, the participant will be asked to temporarily convert his daily dosing to prednisolone/prednisone during a short period of time around RGX-202 administration. He will be allowed to revert back to his baseline vamorolone regimen at the original per kilogram dose at which he entered the study and should remain on this for 24 months unless the investigator determines that this is not clinically indicated or possible.
* Participant has detectable AAV8 total binding antibodies in serum.
* Participant has impaired cardiac function defined as a left ventricular ejection fraction of < 55% on screening cardiac assessments echocardiogram or MRI).
* Participant is not a good candidate for the study, in the opinion of the investigator.

Min Age: 1 Year | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 65 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Part 1 Safety measured by incidence of Adverse Events and Serious Adverse Events | 52 weeks
  Evaluate incidences of AEs and SAEs
Part 2 and 3 Pharmacodynamic | 12 weeks
  Proportion of participants whose RGX-202 microdystrophin protein expression determined in their muscle biopsy is ≥ 10%

SECONDARY OUTCOMES:
Time to Stand (TTSTAND) | 52 Weeks (Part 1); 52 and 104 Weeks (Part 2 &3)
  Values will include time (seconds) and velocity (tasks/second)
Time to Walk/Run 10 meters (TTWR) | 52 Weeks (Part 1) and 104 Weeks (Part 2 &3)
  Values will include time (seconds) and velocity (meters/second)
Time to Climb 4 Stairs (TTCLIMB) | 52 Weeks (Part 1); 52 and 104 Weeks (Part 2 &3)
  Values will include time (seconds) and velocity (tasks/second)
North Star Ambulatory Assessment (NSAA) | 52 Weeks (Part 1) and; 52 and 104 Weeks (Part 2 &3)
  Performance-based assessment of muscle strength and function using a 17-item scale, with all items rated 0,1, or 2, with higher score indicating better performance. The NSAA total score is the sum of the 17 items, ranging from 0 to 34. NSAA linearized score ranges from 0 to 100.
Peabody Developmental Motor Scale, Third Edition (PDMS-3); Body Control Subtest | 52 Weeks (Part 1); 52 and 104 Weeks (Part 2 &3)
  The PDMS-3 is a norm-referenced developmental assessment that measures motor skills of young children. The Body Control subtest measures the child's ability to maintain balance and postural reactions in a variety of positions. Motor skills appropriate for the child's developmental level are administered and rated 0, 1, or 2, with higher score indicating better performance. Body Control subtest total raw scores range from 0 to 112. Age equivalent and scaled scores will also be generated. PDMS-3 Body Control subtests is included for participants age <4 at screening.
Peabody Developmental Motor Scale, Third Edition (PDMS-3); Body Transport Subtest | 52 Weeks (Part 1); 52 and 104 Weeks (Part 2 &3)
  The PDMS-3 is a norm-referenced developmental assessment that measures motor skills of young children. The Body Transport subtest measures the child's ability to move from one place to another, including walking, running, jumping forward, and skipping. Motor skills appropriate for the child's developmental level are administered and rated 0, 1, or 2, with higher score indicating better performance. Body Transport subtest total raw score ranges from 0 to 63. Age equivalent and scaled scores will also be generated. PDMS-3 Body Control subtests is included for participants age <4 at screening.
Part 2 and 3: Stride velocity 95th centile | 104 weeks
  Assessment of peak ambulatory performance captured by wearable activity monitoring device. For velocity measures, higher values indicate greater function.
Part 1 Microdystrophin protein expression | 12 weeks
  RGX-202 microdystrophin protein levels determined in muscle biopsy.
Part 1 Pharmacokinetics (PK) | 12 weeks (muscle) and 52 weeks (serum)
  Vector genome concentrations as measured by polymerase chain reaction [PCR] to RGX-202 deoxyribonucleic acid [DNA] in muscle and serum.
Part 1 Vector Shedding | 52 weeks
  Vector genome concentrations as measured by polymerase chain reaction [PCR] to RGX-202 deoxyribonucleic acid [DNA] in urine.
Part 2 and 3 Microdystrophin protein expression | 12 weeks
  RGX-202 microdystrophin protein levels determined in muscle biopsy.
Part 2 and 3 Safety measured by incidence of Adverse Events and Serious Adverse Events | 104 weeks
  Evaluate incidences of AEs and SAEs
Part 2 and 3 Pharmacokinetics (PK) | 12 weeks (muscle) 52 weeks (serum)
  Vector genome concentrations as measured by polymerase chain reaction [PCR] to RGX-202 deoxyribonucleic acid [DNA] in muscle and serum.
Part 2 and 3 Vector Shedding | 52 weeks
  Vector genome concentrations as measured by polymerase chain reaction [PCR] to RGX-202 deoxyribonucleic acid [DNA] in urine, feces, and saliva.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (13):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Stanford School of Medicine /Division of Neuromuscular Medicine, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Cincinnati Children's, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Hospital of Richmond at Virginia Commonwealth University, Richmond, Virginia
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Children's Hospital London Health Science Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

REFERENCES:
- See also: For additional information on how to participate (or be considered for the study) please follow this link. — https://mytomorrows.com/trials/affinity-duchenne/en-us/?utm_source=ct-gov&utm_medium=referral
- See also: Related Info — http://www.regenxbiodmdtrials.com